CLINICAL TRIAL: NCT06129149
Title: Resources for Resiliency (R4R) Advance Care Planning: A Pilot Study to Test a Trauma-Informed Care-adapted Advance Care Planning Intervention Among Affordable Housing Residents in Nashville
Brief Title: The R4R Advance Care Planning Pilot Study
Acronym: R4RACP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Christine Kimpel, Principal Investigator, Vanderbilt University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 231919
Record Dates: First submitted 2023-11-08; First posted 2023-11-13 (Actual); Results first posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Advance Care Planning
Keywords: advance care planning; affordable housing; housing insecurity; social determinants of health; trauma-informed care; qualitative research; implementation science

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): All participants will participate in this single arm study consisting of three visits: visit 1 (baseline data collection), visit 2 (intervention followed by brief qualitative debrief interview), and visit 3 (30-day follow-up data collection)
  Interventions: Behavioral: Trauma-Informed Care-adapted and Checklist-guided ACP intervention

INTERVENTIONS:
Behavioral: Trauma-Informed Care-adapted and Checklist-guided ACP intervention — The intervention will consist of a single one- to two-hour visit wherein the PI (Kimpel) will facilitate a flexible conversational approach with the resident (and, optionally, a healthcare decision-maker) in a quiet, private location in the resiliency hub. Using a conversation checklist adapted from a narrative synthesis of advance care planning (ACP) guides (Fahner et al., 2019), the PI will explore ACP with participants and use each visit to continually adapt the checklist and approach with trauma-informed care (TIC) principles: safety, trustworthiness and transparency, peer support, collaboration and mutuality, empowerment, and choice, and cultural, historical, and gender issues. Adverse Childhood Experiences and previous death-related experiences assessed during baseline data collection will be used to tailor the discussion to carefully explore relevant history to assess resident ACP values, preferences, and goals.

SUMMARY:
Affordable housing residents continue to experience multi-faceted insecurity and advance care planning (ACP) challenges even after obtaining secure housing, resulting in significant inequities in quality of care during times of cognitive incapacity. To promote proactive planning for affordable housing residents, this proposal is for a pilot study to test a novel trauma-informed care adapted advance care planning intervention with the following aims: to test initial efficacy of the intervention on ACP outcomes (Aim 1) and determine resident perceptions of intervention acceptability, appropriateness, and feasibility and perceived implementation barriers and facilitators (Aim 2). These data will support the development of a larger scale study of ACP interventions within a resiliency-based hub model to comprehensively support whole-person care and proactive planning for times of cognitive incapacity.

DETAILED DESCRIPTION:
Long-term objectives and goals. Vanderbilt University School of Nursing (VUSN) and Urban Housing Solutions (UHS) - the second largest provider of affordable housing in Nashville - are partners with the long-term goal of reducing health disparities among medically-underserved UHS residents in Nashville. This partnership is developing resiliency hubs that will provide essential services and support within a communal setting at the housing facility. Previous literature and data findings support that similar populations to this community lack information about and access to advance care planning (ACP), which specifies their healthcare wishes during cognitive incapacitation or end-of-life, and nationwide research shows significant disparities regarding ACP participation among low-income populations. The short-term goal of the proposed work is to pilot test a Hybrid type 1, single-arm, pre-post intervention to assess the initial efficacy and implementation outcomes of a trauma-informed care (TIC)-adapted ACP intervention to improve learning and communication for times of decisional incapacity among UHS residents, within the context of a resiliency hub model. This is a necessary first step for developing a long-term research portfolio dedicated to addressing ACP disparities and promoting equitable end-of-life planning among low-income, medically-underserved populations.

ELIGIBILITY:
Inclusion Criteria:

* an adult (18+) residing in an affordable housing unit that does not have a completed advance directive

Exclusion Criteria:

* inability to provide informed consent or participate in the intervention due to cognitive, auditory, visual impairment or non-English language barrier

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2024-05-14 (Actual); Primary Completion 2024-12-10 (Actual); Study Completion 2024-12-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kate Clouse, PhD, MPH, Principal Investigator — Vanderbilt University; Christian Ketel, DNP, RN, FNAP, Principal Investigator — Vanderbilt University
Locations (1):
- Urban Housing Solutions, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
Quantitative and qualitative data will be collected during this study. Due to the small size of our sample and the specificity of our recruitment locations, we have developed the following plan to share data while protecting participant privacy. De-identified data will be made available to individuals within Vanderbilt University to promote the research and training of the Vanderbilt community. We will share study materials with researchers outside of the institution, such as the study protocol , SAP, ICF, etc., upon individual request and with institutional permission.
Time Frame: The data will become available 3 months following publication of outcomes and will remain available for at least 5 years
Access Criteria: Data will be made available to researchers who provide a methodologically sound proposal that has been approved by the Vanderbilt Institutional Review Board and the study executive committee.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention
Started | 30
Completed | 29
Not Completed | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Population: One participant died before 30-day follow-up data could be collected, and their data was excluded from the final analysis.
Arm/Group | Intervention
Number analyzed (Participants) | 30
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 60 [56 to 64]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 28
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 17
  White | 11
  More than one race | 2
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Advance Care Planning Values/Beliefs
Description: Advance Care Planning Values/Beliefs Scale, Possible scores: 7-35, Higher summed scores are worse, indicating a higher number of advance care planning misconceptions
Time Frame: Baseline to 30 days
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 29
Score on a scale
  Baseline | 24.9 (6.1)
  30-days post-intervention | 26.3 (4.5)

2. Primary Outcome: Advance Care Planning Processes
Description: Advance Care Planning Processes Scale; Possible scores: 15-75; Higher summed scores are better and indicate higher participation in advance care planning processes
Time Frame: Baseline to 30 days
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 29
Score on a scale
  Baseline | 29.2 (11.9)
  30-days post-intervention | 43.8 (14.4)

3. Primary Outcome: Advance Care Planning Actions
Description: Stages of Change for Advance Care Planning Behaviors Scale; Possible Scores: 0-24; Higher summed scores are better and indicate higher levels of advance care planning participation.
Time Frame: Baseline to 30 days
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 29
Score on a scale
  Baseline | 8.6 (7.0)
  30-days post-intervention | 12.6 (5.9)

4. Primary Outcome: Implementation Acceptability
Description: Acceptability of Intervention Measure: Possible scores: 4-20; Higher scores indicate greater acceptability.
  The result is the percentage of the participants who had a score ≥15 as hypothesized
Time Frame: 30-day post-intervention follow-up (Visit 3)
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention
Number analyzed (Participants) | 29
Participants | 29

5. Primary Outcome: Implementation Appropriateness
Description: Intervention Appropriateness Measure: Possible scores: 4-20; Higher scores indicate greater appropriateness.
  The result is the percentage of the participants who had a score ≥15 as hypothesized
Time Frame: 30-day post-intervention follow-up (Visit 3)
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention
Number analyzed (Participants) | 29
Participants | 24

6. Primary Outcome: Implementation Feasability
Description: Feasibility of Intervention Measure: Possible scores: 4-20; Higher scores indicate greater feasibility.
  The result is the percentage of the participants who had a score ≥15 as hypothesized
Time Frame: 30-day post-intervention follow-up (Visit 3)
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention
Number analyzed (Participants) | 29
Participants | 28

ADVERSE EVENTS:
Time Frame: 7 months
Arm/Group | Intervention
All-Cause Mortality (participants affected / at risk) | 1/30
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 0/30

LIMITATIONS AND CAVEATS:
No comparison group. Nonprobability sampling. No adjusted statistical analysis due to small sample size Single site

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-11-07): https://cdn.clinicaltrials.gov/large-docs/49/NCT06129149/Prot_SAP_002.pdf
  • Informed Consent Form (2024-09-20): https://cdn.clinicaltrials.gov/large-docs/49/NCT06129149/ICF_000.pdf